CLINICAL TRIAL: NCT01720108
Title: Extended Venous Thromboembolism Prophylaxis Comparing Rivaroxaban to Aspirin Following Total Hip and Knee Arthroplasty
Acronym: EPCAT II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: David Anderson (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, David Anderson, Head, Department of Medicine, CDHA, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EPCATII.001
Record Dates: First submitted 2012-10-30; First posted 2012-11-02 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Rivaroxaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rivaroxaban (Active Comparator): rivaroxaban 10mg x 9 days for total knee arthroplasty patients; x 30 days for total hip athroplasty patients
  Interventions: Drug: rivaroxaban and ASA
- ASA (Experimental): ASA 81mg x 9 days for total knee arthroplasty patients; x 30 days for total hip athroplasty patients
  Interventions: Drug: rivaroxaban and ASA

INTERVENTIONS:
Drug: rivaroxaban and ASA

SUMMARY:
In this study the investigators want to look at whether using aspirin instead of rivaroxaban (after initial treatment with rivaroxaban) works as well at preventing blood clots while also reducing risk of bleeding and is more cost effective in patients who have either a total hip replacement or total knee replacement.

ELIGIBILITY:
Inclusion Criteria:

1. All patients undergoing elective total hip or knee arthroplasty at the participating institutions will be potentially eligible for this study

Exclusion Criteria:

1. Hip or lower limb fracture in the previous three months
2. Metastatic cancer
3. Life expectancy less than 6 months
4. History of major bleeding that in the judgment of the investigator precludes use of anticoagulant prophylaxis
5. History of aspirin allergy, active peptic ulcer disease or gastritis that in judgment of investigator precludes use of aspirin
6. History of significant hepatic disease or any other condition that in the judgement of the investigator precludes the use of rivaroxaban
7. Creatinine clearance less than 30 ml per minute
8. Platelet count less than 100 x 109 /L
9. Need for long-term anticoagulation due to a preexisting co-morbid condition or due to the development of venous thromboembolism following surgery but prior to randomization
10. Did not or will not receive rivaroxaban post-operatively for VTE prophylaxis
11. Bilateral total hip arthroplasty or simultaneous hip and knee arthroplasty
12. Major surgical procedure within the previous three months
13. Requirement for major surgery post arthroplasty within 90 day period
14. Chronic daily aspirin use with dose greater than 100 mg a day
15. Women of child bearing potential who are not abstinent or do not use appropriate contraception throughout the study drug period
16. Geographical inaccessibility for follow-up
17. Unwilling or unable to give consent
18. Previous participation in the study
19. Concomitant use with drugs that are strong inhibitors or inducers of both P-gp and CYP3A4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3426 (Actual)
Dates: Start 2013-02-24 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
symptomatic venous thromboembolism | up to 4 years
major or clinically relevant non-major bleeding | up to 4 years

SECONDARY OUTCOMES:
survival | up to 4 years
myocardial infarction | up to 4 years
stroke | up to 4 years
wound infection | up to 4 years
cost-effectiveness | up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: David R Anderson, MD, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Capital Health, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Anderson DR, Dunbar M, Murnaghan J, Kahn SR, Gross P, Forsythe M, Pelet S, Fisher W, Belzile E, Dolan S, Crowther M, Bohm E, MacDonald SJ, Gofton W, Kim P, Zukor D, Pleasance S, Andreou P, Doucette S, Theriault C, Abianui A, Carrier M, Kovacs MJ, Rodger MA, Coyle D, Wells PS, Vendittoli PA. Aspirin or Rivaroxaban for VTE Prophylaxis after Hip or Knee Arthroplasty. N Engl J Med. 2018 Feb 22;378(8):699-707. doi: 10.1056/NEJMoa1712746. PMID 29466159